CLINICAL TRIAL: NCT00910273
Title: Effects of Etanercept on Endothelial Function and Carotid Intima-media Thickness (IMT) in Patients With Active AS
Brief Title: Effects of Etanercept on the Heart, Veins and Thickness of Certain Major Arteries In Ankylosing Spondylitis Patients
Acronym: CREST
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Lincoln Medical and Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0881A3-4458
Record Dates: First submitted 2009-05-27; First posted 2009-05-29 (Estimated); Results first posted 2016-01-13 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2015-12

CONDITIONS: Ankylosing Spondylitis
Keywords: IMT evaluation in AS patients treated with etanercept
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): etanercept 50 mg/week
  Interventions: Drug: etanercept

INTERVENTIONS:
Drug: etanercept — etanercept 50 mg/week
  Other Names: Enbrel

SUMMARY:
Study to assess whether etanercept therapy is able to increase flow-mediated vasodilatation in AS, and whether etanercept can modify the intima-media thickness (IMT) in these patients

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of AS, as defined by Modified New York Criteria for Ankylosing Spondylitis.
2. AS with active disease as defined by Bath Ankylosing Spondylitis Disease Activity Index (BASDAI, see Attachment 4) >= 4 at screening visit.
3. Patients capable, in the opinion of the investigator, of complying with the treatment schedule and doses throughout the 52 weeks
4. Agreement by male subjects who are not surgically sterile and female subjects who are not surgically sterile or postmenopausal to use reliable methods of birth control for the duration of the study.
5. Ability to self-inject drug or have a designee who can do so.
6. Ability to store injectable test article at 2ºC to 8ºC.

Exclusion Criteria:

1. Pregnancy confirmed by test taken at screening in all women except those who were surgically sterile or at least 1 year postmenopausal. Sexually active women of childbearing potential participating in the study must use a medically acceptable form of contraception that needs to be continued for 15 days following discontinuation of the test article.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- Italy (4):
  - Pfizer Investigational Site, Bologna
  - Pfizer Investigational Site, Prato
  - Pfizer Investigational Site, Reggio Emilia
  - Pfizer Investigational Site, Roma

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0881A3-4458&StudyName=Effects%20of%20etanercept%20on%20the%20heart%2C%20veins%20and%20thickness%20of%20certain%20major%20arteries%20In%20Ankylosing%20Spondylitis%20Patients

RESULTS

PARTICIPANT FLOW:
Groups:
- Etanercept: Participants received etanercept (50 milligrams [mg]) subcutaneous (sc) injection once per week for 52 weeks.
- Placebo: Participants received matched placebo sc injection once per week for 52 weeks.
Period: Overall Study
Arm/Group | Etanercept | Placebo
Started | 18 | 16
Completed | 0 | 3
Not Completed | 18 | 13
Not completed — Lack of Efficacy | 6 | 9
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Discontinuation of study by sponsor | 8 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Etanercept | Placebo | Total
Number analyzed (Participants) | 18 | 16 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.47 (8.69) | 46.83 (13.14) | 42.93 (11.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 10 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Flow-Mediated Dilatation (FMD) at Week 12
Description: Brachial artery (BA) FMD equals (=)(maximum diameter minus[-] baseline diameter divided by baseline diameter) times (*) 100 percent (%). Ultrasound images of BA at rest were followed by blood pressure (BP) cuff inflated to at least 50 millimeters of mercury (mm Hg) above participants systolic BP for 5 minutes. Cuff released and reactive hyperaemia was produced. BA was imaged continuously from 30 seconds prior cuff inflation to 2 minutes after cuff deflation. Higher scores indicate improved endothelial function.
Time Frame: Baseline, Week 12
Population: Modified Intent to Treat Population (mITT): all randomized participants who received at least one dose of test article followed by at least one available evaluation; n=number of participants evaluable at specific time point
Measure: Mean (Standard Deviation); unit: percentage of BA diameter
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 17 | 15
percentage of BA diameter
  Baseline (n=17, 15) | 10.09 (5.93) | 13.42 (7.70)
  Change at Week 12 (n=16, 12) | 4.10 (11.41) | 0.25 (7.35)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Null Hypothesis: No difference in Change in FMD at 12 weeks for Etanercept and placebo. Alternative Hypothesis: Difference in Change in FMD at 12 weeks for Etanercept and placebo. Sample size of 36 subjects per treatment arm was planned based on an expected difference of 0.9 in FMD (Standard Deviation [SD] 1.5), with 80% power and 5% significance level; Test type: Superiority or Other; p = 0.608, Mixed Models Analysis; Mean Difference (Final Values) = 1.72, 95% CI 2-sided [-5.14 to 8.58]

2. Secondary Outcome: Change From Baseline in Flow-Mediated Dilatation at Weeks 4, 24, 36, and 52
Description: BA FMD =(maximum diameter -baseline diameter divided by baseline diameter) * 100%. Ultrasound images of BA at rest were followed by BP cuff inflated to at least 50 mm Hg above participants systolic BP for 5 minutes. Cuff released and reactive hyperaemia was produced. BA was imaged continuously from 30 seconds prior cuff inflation to 2 minutes after cuff deflation. Higher scores indicate improved endothelial function. Change: Week x observation minus Baseline observation.
Time Frame: Baseline, Weeks 4, 24, 36, and 52 or Early Termination (ET)
Population: mITT; n=number of participants evaluable at specific time point
Measure: Mean (Standard Deviation); unit: percentage of BA diameter
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 17 | 15
percentage of BA diameter
  Change at Week 4 (n=17, 13) | 2.56 (9.51) | -0.68 (4.75)
  Change at Week 24 (n=9, 4) | 3.89 (10.56) | 3.20 (5.75)
  Change at Week 36 (n=7, 4) | 6.24 (5.53) | 5.18 (7.33)
  Change at Week 52 (n=4, 3) | 8.14 (5.65) | 12.13 (5.28)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Week 4; Test type: Superiority or Other; p = 0.476, Mixed Models Analysis; Mean Difference (Final Values) = 1.82, 95% CI 2-sided [-3.35 to 7.00] — Analyses available for Week 4 only, due to limited number of participants for Week 24 to Week 52

3. Secondary Outcome: Change From Baseline in Carotid Intima Media Thickness (IMT) at Weeks 12 and 52
Description: Change in IMT in the distal common carotid arteries (CCA), common bulbs (CB), and internal carotid arteries (ICA) as determined by ultrasound. Higher scores indicate worsening in cardiovascular risk assessment. Change: Week x observation minus Baseline observation.
Time Frame: Baseline, Week 12 and 52 or ET
Population: mITT; n=number of participants evaluable at specific time point; N=number of participants evaluable
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 17 | 14
mm
  CCA Baseline (n=17, 14) | 0.65 (0.20) | 0.77 (0.13)
  CCA Change at Week 12 (n=16, 11) | 0.00 (0.15) | -0.09 (0.16)
  CCA Change at Week 52 (n=4, 2) | 0.00 (0.08) | 0.08 (0.01)
  CB Baseline (n=17, 14) | 0.76 (0.16) | 0.89 (0.17)
  CB Change at Week 12 (n=16, 11) | -0.03 (0.11) | -0.02 (0.12)
  CB Change at Week 52 (n=4, 2) | -0.05 (0.19) | 0.03 (0.46)
  ICA Baseline (n=17, 14) | 0.67 (0.19) | 0.75 (0.32)
  ICA Change at Week 12 (n=16, 11) | -0.03 (0.16) | -0.07 (0.28)
  ICA Change at Week 52 (n=4, 2) | -0.03 (0.19) | -0.27 (0.90)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Week 12; Common Carotid Artery; Due to limited number of participants with visits after Week 12 analysis limited to Week 12; Test type: Superiority or Other; p = 0.650, ANCOVA; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.08 to 0.13]
Statistical Analysis 2: Comparison: Etanercept vs Placebo; Week 12; Common Bulb; Due to limited number of participants with visits after Week 12 analysis limited to Week 12; Test type: Superiority or Other; p = 0.513, ANCOVA; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.13 to 0.07]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; Week 12; Internal Carotid Artery; Due to limited number of participants with visits after Week 12 analysis limited to Week 12; Test type: Superiority or Other; p = 0.592, ANCOVA; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.14 to 0.08]

4. Secondary Outcome: Change From Baseline Lipid Parameters at Weeks 4, 12, 24, 36 and 52
Description: Mean Total Cholesterol (TC), Low Density Lipoprotein (LDL) and Triglyceride (TGL) blood concentrations, lower values indicated improvement in cardiovascular risk. Mean High Density Lipoprotein (HDL), higher values indicated improvement in cardiovascular risk. Change: Week x observation minus Baseline observation. Baseline value was used when present, otherwise valid screening value used as baseline if within 14 days of first test article injection.
Time Frame: Baseline, Weeks 4, 12, 24, 36 and 52 or ET
Population: mITT; n=number of participants evaluable at specific time point; N=number of participants evaluable
Measure: Mean (Standard Deviation); unit: millimole/Liter (mmol/L)
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 16 | 15
millimole/Liter (mmol/L)
  TC Baseline (n=16, 15) | 4.39 (0.97) | 4.53 (0.92)
  TC Change at Week 4 (n=16, 13) | 0.25 (0.61) | -0.16 (0.96)
  TC Change at Week 12 (n=15, 12) | 0.30 (0.60) | -0.06 (0.64)
  TC Change at Week 24 (n=9, 4) | 0.27 (0.61) | 0.14 (0.29)
  TC Change at Week 36 (n=7, 4) | 0.50 (0.61) | 0.03 (0.49)
  TC Change at Week 52 (n=4, 3) | -0.06 (0.55) | 0.14 (0.50)
  LDL Baseline (n=16, 15) | 2.76 (1.25) | 3.02 (1.00)
  LDL Change at Week 4 (n=15, 12) | 0.08 (0.62) | 0.08 (0.55)
  LDL Change at Week 12 (n=15, 12) | 0.27 (1.34) | 0.03 (0.39)
  LDL Change at Week 24 (n=9, 4) | 0.04 (0.40) | 0.34 (0.50)
  LDL Change at Week 36 (n=7, 4) | 0.22 (0.48) | -0.01 (0.99)
  LDL Change at Week 52 (n=4, 3) | -0.82 (0.96) | 0.46 (0.86)
  HDL Baseline (n=16, 15) | 1.29 (0.63) | 1.18 (0.32)
  HDL Change at Week 4 (n=15, 12) | 0.10 (0.28) | -0.00 (0.14)
  HDL Change at Week 12 (n=15, 12) | 0.07 (0.19) | -0.03 (0.16)
  HDL Change at Week 24 (n=9, 4) | 0.11 (0.26) | 0.08 (0.15)
  HDL Change at Week 36 (n=7, 4) | 0.19 (0.21) | 0.30 (0.54)
  HDL Change at Week 52 (n=4, 3) | -0.01 (0.24) | -0.02 (0.23)
  TGL Baseline (n=16, 15) | 0.96 (0.54) | 1.25 (0.67)
  TGL Change at Week 4 (n=15, 12) | 0.14 (0.33) | -0.06 (0.65)
  TGL Change at Week 12 (n=15, 12) | 0.20 (0.50) | -0.12 (0.71)
  TGL Change at Week 24 (n=9, 4) | 0.24 (0.56) | -0.91 (0.83)
  TGL Change at Week 36 (n=7, 4) | 0.33 (0.50) | -0.76 (0.43)
  TGL Change at Week 52 (n=4, 3) | 0.45 (0.63) | -0.99 (0.82)

5. Secondary Outcome: Change From Baseline in Total Serum Homocysteine at Weeks 4, 12, 24, 36 and 52
Description: Mean serum homocysteine blood concentrations. Lower values of homocysteine indicate improvement in inflammation. Change: Week x observation minus Baseline observation. Baseline value was used when present, otherwise valid screening value used as baseline if within 14 days of first test article injection.
Time Frame: Baseline, Weeks 4, 12, 24, 36 and 52 or ET
Population: mITT; n= number of participants evaluable at specific time point; N=number of participants evaluable
Measure: Mean (Standard Deviation); unit: micromole/liter (µmol/L)
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 16 | 15
micromole/liter (µmol/L)
  Baseline (n=16, 15) | 11.31 (4.18) | 14.59 (9.63)
  Change at Week 4 (n=15, 11) | 0.31 (3.16) | 0.33 (4.13)
  Change at Week 12 (n=15, 12) | -0.07 (2.51) | 0.13 (4.05)
  Change at Week 24 (n=8, 4) | -1.72 (3.52) | -1.40 (10.40)
  Change at Week 36 (n=7, 4) | 1.65 (1.92) | -2.58 (8.05)
  Change at Week 52 (n=4, 3) | 1.49 (2.20) | -6.98 (10.79)

6. Secondary Outcome: Change From Baseline in Erythrocyte Sedimentation Rate (ESR) at Weeks 4, 12, 24, 36 and 52
Description: ESR is a laboratory test that provides a non-specific measure of inflammation. The test assesses the rate at which red blood cells fall in a test tube. Normal range is 0-30 mm/hour (hr). A higher rate is consistent with inflammation. Change: Week x observation minus Baseline observation. Baseline value was used when present, otherwise valid screening value used as baseline if within 14 days of first test article injection.
Time Frame: Baseline, Weeks 4, 12, 24, 36 and 52 or ET
Population: mITT; N=number of participants evaluable; n= number of participants evaluable at specific time point
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 16 | 15
mm/hr
  Baseline (n=16, 15) | 42.85 (37.73) | 45.80 (42.50)
  Change at Week 4 (n=16, 13) | -21.49 (28.82) | -1.25 (27.53)
  Change at Week 12 (n=15, 12) | -29.47 (36.84) | 4.40 (17.39)
  Change at Week 24 (n=9, 4) | -31.89 (28.62) | 4.73 (15.60)
  Change at Week 36 (n=7, 4) | -31.06 (25.13) | -3.62 (4.30)
  Change at Week 52 (n=5, 3) | -37.47 (23.66) | -6.15 (7.52)

7. Secondary Outcome: Change From Baseline in C-Reactive Protein (CRP) at Weeks 4, 12, 24, 36, 52
Description: CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement. Change: Week x observation minus Baseline observation. Baseline value was used when present, otherwise valid screening value used as baseline if within 14 days of first test article injection.
Time Frame: Baseline, Weeks 4, 12, 24, 36 and 52 or ET
Population: mITT; N=number of participants evaluable; n= number of participants evaluable at specific time point
Measure: Mean (Standard Deviation); unit: mg/liter (mg/L)
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 16 | 15
mg/liter (mg/L)
  Baseline (n=16, 15) | 19.66 (31.66) | 11.83 (24.64)
  Change at Week 4 (n=15, 13) | -17.46 (30.80) | -1.32 (8.19)
  Change at Week 12 (n=14, 12) | -11.84 (19.45) | 2.01 (6.17)
  Change at Week 24 (n=9, 4) | -25.58 (38.08) | -2.55 (6.45)
  Change at Week 36 (n=7, 4) | -20.96 (37.81) | -3.05 (5.33)
  Change at Week 52 (n=5, 3) | -20.09 (31.74) | -3.58 (6.42)

8. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at Week 4, 12, 24, 36 and 52
Description: BASDAI a validated self assessment tool to determine disease activity in participant with Ankylosing Spondylitis (AS) using a Visual Analog Scale (VAS) of 0 (none) to 10 (very severe) centimeter (cm). Participant answered 6 questions measuring discomfort, pain and fatigue. Final BASDAI score averages the individual assessments for a final score range of 0-10. Change: Week x observation minus Baseline observation. Higher score indicates greater disability. Baseline value was used when present, otherwise valid screening value used as baseline if within 14 days of first test article injection.
Time Frame: Baseline, Weeks 4, 12, 24, 36, and 52 or ET
Population: mITT; n= number of participants evaluable at specific time point
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 17 | 15
Units on a scale
  Baseline (n= 17,15) | 6.21 (1.63) | 6.30 (1.40)
  Change at Week 4 (n=17, 14) | -1.79 (1.81) | -0.10 (1.63)
  Change at Week 12 (n=16, 13) | -3.19 (2.34) | -1.31 (2.56)
  Change at Week 24 (n=9, 4) | -3.86 (1.30) | -5.28 (1.09)
  Change at Week 36 (n=8, 4) | -4.05 (1.47) | -3.06 (3.94)
  Change at Week 52 (n=5, 2) | -4.49 (0.96) | -5.12 (2.07)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Week 4; Test type: Superiority or Other; p = 0.008, Mixed Models Analysis; Mean Difference (Final Values) = -1.77, 95% CI 2-sided [-3.05 to -0.50] — Adjusted mean difference (Etanercept-Placebo)
Statistical Analysis 2: Comparison: Etanercept vs Placebo; Week 12; Test type: Superiority or Other; p = 0.021, Mixed Models Analysis; Mean Difference (Final Values) = -2.02, 95% CI 2-sided [-3.70 to -0.33] — Adjusted mean difference (Etanercept-Placebo)

9. Secondary Outcome: Percentage of Participants With BASDAI 50 Percent (%) Improvement at Weeks 4, 12, 24, 36, and 52
Description: BASDAI a validated self assessment tool used to determine disease activity in participants with AS. Utilizing a VAS of 0 (none) to 10 cm (very severe), participant's answered 6 questions measuring discomfort, pain and fatigue. BASDAI 50 response defined as at least a 50% improvement (decrease) from baseline in BASDAI. Baseline score - score at observation divided by Baseline score * 100 = greater than or equal to 50%.
Time Frame: Weeks 4, 12, 24, 36, and 52 or ET
Population: mITT; N=number of participants evaluable; n=number of participants evaluable at specific time point
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 17 | 14
percentage of participants
  Week 4 (n= 17, 14) | 29.4 | 0
  Week 12 (n=16, 13) | 62.5 | 23.1
  Week 24 (n=9, 4) | 77.8 | 100
  Week 36 (n=8, 4) | 87.5 | 75.0
  Week 52 (n=5, 2) | 80.0 | 100

10. Secondary Outcome: Percentage of Participants With Assessment in Ankylosing Spondylitis (ASAS) 20 at Weeks 4, 12, 24, 36, and 52
Description: ASAS measures symptomatic improvement in Ankylosing Spondylitis (AS) participants ASAS = 4 domains: participant global assessment of disease activity, pain, function, inflammation. ASAS 20 = 20% improvement from baseline and an absolute change greater than or equal to (≥) 10 units on a 0-100 millimeter (mm) scale (0 mm = no disease activity; 100 mm = high disease activity) for ≥ 3 domains, and no worsening in remaining domain.
Time Frame: Week 4, 12, 24, 36, and 52 or ET
Population: mITT; N=number of participants evaluable; n=number of participants evaluable at specific time point
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 17 | 14
percentage of participants
  Week 4 (n=17, 14) | 41.2 | 0
  Week 12 (n=16, 13) | 68.8 | 46.2
  Week 24 (n=9, 4) | 88.9 | 100
  Week 36 (n=8, 4) | 87.5 | 75.0
  Week 52 (n=5, 2) | 100 | 100

11. Secondary Outcome: Percentage of Participants With ASAS 40 at Weeks 4, 12, 24, 36, and 52
Description: ASAS measures symptomatic improvement in Ankylosing Spondylitis (AS) participants ASAS = 4 domains: participant global assessment of disease activity, pain, function, inflammation. ASAS 40 = 40% improvement from baseline and an absolute change ≥ 20 units on a 0-100 mm scale (0 mm = no disease activity, 100 mm = high disease activity) for ≥ 3 domains, and no worsening in remaining domain.
Time Frame: Weeks 4, 12, 24, 36, and 52 or ET
Population: mITT; N=number of participants evaluable; n=number of participants evaluable at specific time point
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 17 | 14
percentage of participants
  Week 4 (n=17, 14) | 29.4 | 0
  Week 12 (n=16, 13) | 56.3 | 38.5
  Week 24 (n=9, 4) | 88.9 | 75.0
  Week 36 (n=8, 4) | 75.0 | 75.0
  Week 52 (n=5, 2) | 100 | 100

12. Secondary Outcome: Percentage of Participants With ASAS 50 at Weeks 4, 12, 24, 36, and 52
Description: ASAS measures symptomatic improvement in Ankylosing Spondylitis (AS) participants ASAS = 4 domains: participant global assessment of disease activity, pain, function, inflammation. ASAS 50 = 50% improvement (vs. baseline) and an absolute change ≥ 20 units on a 0-100 mm scale (0 mm = no disease activity, 100 mm = high disease activity) for ≥ 3 domains, and no worsening in remaining domain.
Time Frame: Weeks 4, 12, 24, 36 and 52 or ET
Population: mITT; N=number of participants with evaluable; n=number of participants evaluable at specific time point
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 17 | 14
percentage of participants
  Week 4 (n=17, 14) | 29.4 | 0
  Week 12 (n=16, 13) | 56.3 | 23.1
  Week 24 (n=9, 4) | 77.8 | 75.0
  Week 36 (n=8, 4) | 75.0 | 75.0
  Week 52 (n=5, 2) | 100 | 100

13. Secondary Outcome: Percentage of Participants With ASAS 70 at Weeks 4, 12, 24, 36, and 52
Description: ASAS measures symptomatic improvement in Ankylosing Spondylitis (AS) participants ASAS = 4 domains: participant global assessment of disease activity, pain, function, inflammation. ASAS 70 = 70% improvement (vs. baseline) and an absolute change ≥ 20 units on a 0-100 mm scale (0 mm = no disease activity, 100 mm = high disease activity) for ≥ 3 domains, and no worsening in remaining domain.
Time Frame: Weeks 4, 12, 24, 36 and 52 or ET
Population: mITT; N=number of participants evaluable; n=number of participants evaluable at specific time point
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 17 | 14
percentage of participants
  Week 4 (n=17, 14) | 11.8 | 0
  Week 12 (n=16, 13) | 25.0 | 7.7
  Week 24 (n=9, 4) | 44.4 | 50.0
  Week 36 (n=8, 4) | 37.5 | 50.0
  Week 52 (n=5, 2) | 40.0 | 50.0

14. Secondary Outcome: Percentage of Participants With ASAS 5/6 at Weeks 4, 12, 24, 36, and 52
Description: ASAS 5/6 consists of 6 domains: the 4 used in ASAS 20 (participant global assessment of disease activity, pain, function, inflammation measured on a 0-100 scale, where 0 = no disease activity and 100=high disease activity) plus spinal mobility and an acute phase reactant, C Reactive Protein (CRP). Achieving ASAS 5/6 requires a 20% improvement compared to baseline in ≥ 5 domains and no worsening in the remaining domain.
Time Frame: Weeks 4, 12, 24, 36 and 52 or ET
Population: mITT; N=number of participants evaluable; n=number of participants evaluable at specific time point
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 17 | 14
percentage of participants
  Week 4 (n=17, 14) | 5.9 | 0
  Week 12 (n=16, 13) | 25.0 | 0
  Week 24 (n=9, 4) | 22.2 | 25.0
  Week 36 (n=8, 4) | 25.0 | 50.0
  Week 52 (n=5, 2) | 40.0 | 50.0

15. Secondary Outcome: Percentage of Participants With ASAS Partial Remission at Weeks 4, 12, 24, 36, and 52
Description: Partial remission defined as a score of less than 20 units (on a scale of 0-100, where 0 = no disease activity and 100 = high disease activity) in each of the 4 Assessment in Ankylosing Spondylitis (ASAS) domains: participant global assessment of disease activity, pain, function, and inflammation. For scale, 100=high disease activity.
Time Frame: Weeks 4, 12, 24, 36 and 52 or ET
Population: mITT; N=number of participants evaluable; n=number of participants evaluable at specific time point
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 17 | 14
percentage of participants
  Week 4 (n=17, 14) | 29.4 | 0
  Week 12 (n=15, 13) | 46.7 | 38.5
  Week 24 (n=8, 4) | 87.5 | 75.0
  Week 36 (n=7, 4) | 71.4 | 75.0
  Week 52 (n=4, 2) | 75.0 | 100

16. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Metrology Index (BASMI) at Week 4, 12, 24, 36, and 52
Description: BASMI is an objective measure of spinal mobility. The BASMI score is composed of 5 measures: cervical rotation, intermalleolar distance, modified Schober's test, lateral flexion and tragus to wall distance. Each measure was scored 0-2 (0=normal mobility, 2=severe reduction) to give a final score ranging 0 to 10. Lower score indicated better spinal mobility. Change: Week x observation minus Baseline observation. Baseline value was used when present, otherwise valid screening value used as baseline if within 14 days of first test article injection.
Time Frame: Baseline, Weeks 4, 12, 24, 36 and 52 or ET
Population: mITT; n=number of participants evaluable at specific time point
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 17 | 15
Units on a scale
  Baseline (n=17, 15) | 3.47 (2.21) | 3.98 (2.48)
  Change at Week 4 (n=17, 14) | -0.41 (0.91) | 0.63 (0.93)
  Change at Week 12 (n=16, 12) | -0.73 (1.23) | 0.15 (1.06)
  Change at Week 24 (n=9, 4) | -0.50 (1.06) | -0.75 (0.96)
  Change at Week 36 (n=8, 4) | -0.88 (1.13) | -0.81 (0.55)
  Change at Week 52 (n=5, 3) | -0.35 (1.58) | -0.75 (0.66)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Week 4; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis; Mean Difference (Final Values) = -1.07, 95% CI 2-sided [-1.74 to -0.40] — Adjusted mean difference (Etanercept-Placebo)
Statistical Analysis 2: Comparison: Etanercept vs Placebo; Week 12; Test type: Superiority or Other; p = 0.029, Mixed Models Analysis; Mean Difference (Final Values) = -0.91, 95% CI 2-sided [-1.72 to -0.10] — Adjusted mean difference (Etanercept-Placebo)

17. Secondary Outcome: Change From Baseline in BASMI-Cervical Rotation at Weeks 4, 12, 24, 36 and 52
Description: While in a neutral position, the participant turned the head as far as possible to the right and then to the left. Using a goniometer the degrees of movement were measured. Two measurements on the right and 2 on the left were made. The best of the two measurements for each side (corresponding to the highest value), were then averaged. Higher score indicated greater spinal mobility. Actual rotation ranged from 3.0 to 99.0 degrees. Change: Week x observation minus Baseline observation. Baseline value was used when present, otherwise valid screening value used as baseline if within 14 days of first test article injection.
Time Frame: Baseline, Weeks 4, 12, 24, 36, 52 or ET
Population: mITT; n= number of participants evaluable at specific time point
Measure: Mean (Standard Deviation); unit: degrees of movement
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 17 | 15
degrees of movement
  Baseline (n= 17, 15) | 57.09 (23.30) | 54.80 (15.31)
  Change at Week 4 (n=17, 14) | 3.79 (9.37) | -2.61 (4.15)
  Change at Week 12 (n=16, 12) | 4.97 (11.04) | -2.79 (6.23)
  Change at Week 24 (n=9, 4) | 4.67 (19.09) | 1.88 (2.59)
  Change at Week 36 (n=8, 4) | 6.50 (18.94) | 7.50 (8.35)
  Change at Week 52 (n=5, 3) | 9.30 (17.09) | 9.17 (9.41)

18. Secondary Outcome: Change From Baseline in BASMI-Intermalleolar Distance at Weeks 4, 12, 24, 36 and 52
Description: Measurement in cm of the distance between the medial malleoli when participant was lying supine with knees straight and feet pointed straight up with legs separated as far as possible, 2 attempts were measured. The best of the two measurements which corresponds to the highest value were reported. Higher score indicated greater spinal mobility. Change: Week x observation minus Baseline observation. Baseline value was used when present, otherwise valid screening value used as baseline if within 14 days of first test article injection.
Time Frame: Baseline, Weeks 4, 12, 24, 36 and 52 or ET
Population: mITT; n= number of participants evaluable at specific time point
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 17 | 15
cm
  Baseline (n= 17, 15) | 103.02 (17.46) | 94.69 (15.38)
  Change at Week 4 (n=17, 14) | -0.34 (9.58) | -4.21 (8.12)
  Change at Week 12 (n=16, 12) | 2.01 (12.78) | 0.90 (7.17)
  Change at Week 24 (n=9, 4) | -0.54 (13.09) | 0.13 (1.75)
  Change at Week 36 (n=8, 4) | 2.14 (13.18) | -2.50 (8.69)
  Change at Week 52 (n=5, 3) | 2.46 (21.22) | 1.33 (1.15)

19. Secondary Outcome: Change From Baseline in BASMI-Modified Schober's Test at Weeks 4, 12, 24, 36 and 52
Description: Measurement in cm of distance between marks originally placed while participant was standing erect 10 cm above and 5 cm below the midpoint of a line that joins the posterior superior iliac spines. Distance between marks was re-measured with participant maximally bent forward, knees fully extended, with supine in full flexion. The measurement was carried out two times and best of the two measurements which corresponds to the highest value were reported. Higher score indicated greater spinal mobility. Change: Week x observation minus Baseline observation. Baseline value was used when present, otherwise valid screening value used as baseline if within 14 days of first test article injection.
Time Frame: Baseline, Weeks 4, 12, 24, 36 and 52 or ET
Population: mITT; n= number of participants evaluable at specific time point
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 17 | 15
cm
  Baseline (n= 17, 15) | 5.00 (4.31) | 4.77 (4.54)
  Change at Week 4 (n=17, 14) | 0.38 (0.78) | 0.11 (0.82)
  Change at Week 12 (n=16, 12) | 1.23 (3.02) | -0.02 (0.86)
  Change at Week 24 (n=9, 4) | 1.41 (3.79) | 0.10 (0.34)
  Change at Week 36 (n=8, 4) | 1.39 (3.88) | -0.05 (0.53)
  Change at Week 52 (n=5, 3) | 2.48 (4.51) | 0.07 (0.40)

20. Secondary Outcome: Change From Baseline in BASMI-Tragus to Wall Distance at Weeks 4, 12, 24, 36 and 52
Description: Measurement in cm of distance between the tragus and wall from the right and left side while participant was standing with back against the wall; knees straight; scapulae, buttocks, and heels against the wall; with head in a neutral position. Two measurements on the right and 2 on the left were made. The best of the two measurements for each side (corresponding to the smallest value), were then averaged. Higher score indicated greater spinal mobility. Change: Week x observation minus Baseline observation. Baseline value was used when present, otherwise valid screening value used as baseline if within 14 days of first test article injection.
Time Frame: Baseline, Weeks 4, 12, 24, 36 and 52 or ET
Population: mITT; n= number of participants evaluable at specific time point
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 17 | 15
cm
  Baseline (n= 17, 15) | 14.31 (2.74) | 14.91 (5.49)
  Change at Week 4 (n=17, 14) | -0.01 (0.82) | 0.43 (0.92)
  Change at Week 12(n=16, 12) | -0.18 (0.90) | -0.33 (0.81)
  Change at Week 24 (n=9, 4) | -0.58 (0.65) | -0.36 (0.82)
  Change at Week 36 (n=8, 4) | -0.26 (1.00) | -0.31 (0.80)
  Change at Week 52 (n=5, 3) | 0.55 (2.67) | -0.10 (0.36)

21. Secondary Outcome: Change From Baseline in BASMI-Lateral Flexion at Weeks 4, 12, 24, 36 and 52
Description: Measurement in cm of distance between participant's middle fingertip and the floor after bending sideways, without bending knees or lifting heels, while attempting to keep shoulders in same place (flexion position). Two measurements on the right and 2 on the left were made. The best of the two measurements for each side (corresponding to the highest value), were then averaged. Higher score indicated greater spinal mobility. Change: Week x observation minus Baseline observation. Baseline value was used when present, otherwise valid screening value used as baseline if within 14 days of first test article injection.
Time Frame: Baseline, Weeks 4, 12, 24, 36 and 52 or ET
Population: mITT; n= number of participants evaluable at specific time point
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 17 | 15
cm
  Baseline (n= 17, 15) | 10.25 (6.25) | 8.00 (6.32)
  Change at Week 4 (n=17, 14) | 0.54 (1.48) | 0.33 (2.46)
  Change at Week 12(n=16, 12) | 0.09 (3.40) | 0.48 (3.78)
  Change at Week 24 (n=9, 4) | 3.01 (3.77) | 0.31 (0.58)
  Change at Week 36 (n=8, 4) | 2.06 (2.35) | -0.69 (1.25)
  Change at Week 52 (n=5, 3) | 2.38 (2.84) | -0.80 (1.63)

22. Secondary Outcome: Change From Baseline in Occiput-to-Wall Distance at Weeks 4, 12, 24, 36 and 52
Description: While participant stood with back against the wall and during maximal effort to touch head to the wall, the distance between the occiput (back of head) and the wall was measured. The measurement of two attempts was made and best of the two measurements which corresponds to the highest value were reported. Lower scores indicated improvement in spinal mobility. Change: Week x observation minus Baseline observation. Baseline value was used when present, otherwise valid screening value used as baseline if within 14 days of first test article injection.
Time Frame: Baseline, Weeks 4, 12, 24, 36 and 52 or ET
Population: mITT; n= number of participants evaluable at specific time point
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 17 | 15
cm
  Baseline (n=17, 15) | 7.67 (3.98) | 9.77 (5.71)
  Change at Week 4 (n=17, 14) | -0.13 (0.88) | 0.89 (1.82)
  Change at Week 12 (n=16, 12) | -0.44 (1.11) | 0.53 (2.00)
  Change at Week 24 (n=9, 4) | -0.14 (1.89) | 0.18 (0.71)
  Change at Week 36 (n=8, 4) | 0.78 (2.06) | -0.40 (1.77)
  Change at Week 52 (n=5, 3) | -0.24 (1.64) | -1.17 (1.61)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Week 4; Test type: Superiority or Other; p = 0.041, Mixed Models Analysis; Mean Difference (Final Values) = -1.09, 95% CI 2-sided [-2.13 to -0.05] — Adjusted mean difference (Etanercept-Placebo)
Statistical Analysis 2: Comparison: Etanercept vs Placebo; Week 12; Test type: Superiority or Other; p = 0.048, Mixed Models Analysis; Mean Difference (Final Values) = -1.28, 95% CI 2-sided [-2.55 to -0.01] — Adjusted mean difference (Etanercept-Placebo)

23. Secondary Outcome: Change From Baseline in Chest Expansion at Weeks 4, 12, 24, 36 and 52
Description: Chest expansion defined as the difference in thoracic circumference during full expiration versus full inspiration, measured in cm at the fourth intercostal space (nipple line) while participant was standing. Measurement taken twice and best of the two measurements (corresponding to the highest value of inspiration and smallest value for expiration), were then averaged. Greater chest circumference indicated improvement in spinal mobility. Change: Week x observation minus Baseline observation. Baseline value was used when present, otherwise valid screening value used as baseline if within 14 days of first test article injection.
Time Frame: Baseline, Weeks 4, 12, 24, 36 and 52 or ET
Population: mITT; n= number of participants evaluable at specific time point; Due to limited number of participants with visits after Week 12 analysis limited to Week 12
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 17 | 15
cm
  Baseline (n=17, 15) | 4.75 (2.19) | 4.50 (1.75)
  Change at Week 4 (n=17, 14) | -0.33 (2.70) | -0.42 (1.00)
  Change at Week 12 (n=16, 12) | 0.22 (3.00) | -0.37 (1.53)
  Change at Week 24 (n=9, 4) | 0.68 (1.86) | -0.73 (1.55)
  Change at Week 36 (n=8, 4) | 0.31 (1.50) | -0.60 (1.78)
  Change at Week 52 (n=5, 3) | 0.58 (1.70) | -0.13 (2.73)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Week 4; Test type: Superiority or Other; p = 0.575, Mixed Models Analysis; Mean Difference (Final Values) = 0.34, 95% CI 2-sided [-0.89 to 1.57] — Adjusted mean difference (Etanercept-Placebo)
Statistical Analysis 2: Comparison: Etanercept vs Placebo; Week 12; Test type: Superiority or Other; p = 0.204, Mixed Models Analysis; Mean Difference (Final Values) = 0.89, 95% CI 2-sided [-0.52 to 2.30] — Adjusted mean difference (Etanercept-Placebo)

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Etanercept | Placebo
Serious Adverse Events (participants affected / at risk) | 1/18 | 0/16
Other Adverse Events (participants affected / at risk) | 9/18 | 3/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=18) | Placebo (N=16)
Renal mass (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=18) | Placebo (N=16)
Tooth abscess (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 1 | 0
Febrile infection (Infections and infestations) | 1 | 0
Injection site erythema (General disorders) | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Due to early termination and few participants attending visits after Week 12, statistical analysis limited to Week 12.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.